CLINICAL TRIAL: NCT07259356
Title: Effect of Blood Flow Restriction Training on the Subjective Perception of Pain in Hemophilic Arthropathy of the Knee Joint
Brief Title: Feasibility and Safety of Blood-Flow-Restriction Training in Patients With Hemophilia
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Alexander Franz, Prinicipal Investigator, University Hospital, Bonn
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2024_H
Record Dates: First submitted 2025-05-13; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-05

CONDITIONS: Hemophilia
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Condition (Active Comparator): Sham-BFR Leg Press Exercise
  Interventions: Device: Control
- Intervention Condition (Experimental): BFR Leg Press Exercise
  Interventions: Device: BFR Exercise (50% of the LOP) while Leg Press Exercise (4 Sets, All out)

INTERVENTIONS:
Device: Control — Sham-BFR Exercise (20mmHg) while Leg Press Exercise (4 Sets, All out)
  Arms: Control Condition
Device: BFR Exercise (50% of the LOP) while Leg Press Exercise (4 Sets, All out) — BFR Exercise (50% of the LOP) while Leg Press Exercise (4 Sets, All out)
  Arms: Intervention Condition

SUMMARY:
In the course of a cross-over study design, 12 patients with hemophilic arthropathy will perform a training load on the knee extensor muscles. The subjects will each perform one intervention with blood flow restriction and one with a Sham-BFR intervention.

ELIGIBILITY:
Inclusion Criteria:

* patients with haemophilia
* Ability for an exercise intervention

Exclusion Criteria:

* Sickle Cell Anemia
* Intravascular stents/bypasses
* Open Wounds/Infections of the lower extremity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Pain threshold | Pre- (Baseline, before Exercise) to immediately Post-Intervention (after the exercise training intervention) and 24 hours after intervention
  Pain threshold measurement (PTT): The test determines the amount of pressure (in kg) over a given area in which a steadily increasing nonpainful pressure stimulus turns into a painful pressure sensation.
Quality of Life Score | Pre- (Baseline, before Exercise) to immediately Post-Intervention (after the exercise training intervention) and 24 hours after intervention
  Hemophilia Joint Health Score

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Bonn, Bonn, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No